CLINICAL TRIAL: NCT04077567
Title: An Extension Study of TS-152 in Subjects with Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS152-3002-JA
Record Dates: First submitted 2019-08-29; First posted 2019-09-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TS-152 30mg SC (Experimental): TS-152 30mg subcutaneously (SC) every 4 weeks
  Interventions: Drug: TS-152
- TS-152 80mg SC (Experimental): TS-152 80mg subcutaneously (SC) every 4 weeks
  Interventions: Drug: TS-152

INTERVENTIONS:
Drug: TS-152 — 30mg,80mg
  Other Names: ozoralizumab

SUMMARY:
To evaluate the long-term safety and efficacy of TS-152 in subjects with Rheumatoid Arthritis who have completed the previous study (TS152-3000-JA study or TS152-3001-JA study).

ELIGIBILITY:
Inclusion Criteria:

1. At visit1(-4 weeks), Subject must be fully informed about the study and must obtain written informed consent from the subject himself.
2. At Visit2(0 week), Subjects must have completed the previous study (TS152-3000-JA or TS152-3001-JA) ,and must have completed all evaluations required at the follow-up visit.

etc.

Exclusion Criteria:

1. Subjects who had serious adverse drug reactions in the previous study.
2. At Visit1(-4 weeks) or Visit2 (0 week), Subjects who have not recovered from clinically important adverse events.

etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | through study completion, an average of 3 year
  To evaluate the Long-term safety of TS-152 in RA patients by incidence of adverse events which include vital signs, and clinical laboratory parameters.
ACR20 | through study completion, an average of 3 year
  Percentage of Subjects who meet the American College of Rheumatology 20% (ACR20) Criteria from baseline of previous study (TS152-3001-JA or TS152-3001-JA).

CONTACTS AND LOCATIONS:
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanaka Y, Miyazaki Y, Kawanishi M, Yamasaki H, Takeuchi T. Long-term safety and efficacy of anti-TNF multivalent VHH antibodies ozoralizumab in patients with rheumatoid arthritis. RMD Open. 2024 Aug 22;10(3):e004480. doi: 10.1136/rmdopen-2024-004480. PMID 39179257